CLINICAL TRIAL: NCT00406029
Title: A Phase 2, 12-Week, Double-Blind, Dose-Finding, Placebo-Controlled Study to Assess the Efficacy and Safety of a Range of SCH 420814 Doses in Subjects With Moderate to Severe Parkinson's Disease Experiencing Motor Fluctuations and Dyskinesias
Brief Title: Dyskinesia in Parkinson's Disease (Study P04501)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04501; MK-3814-013 (Other: Merck)
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease; Movement Disorders; Central Nervous System Diseases; Neurodegenerative Diseases; Brain Diseases
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Central Nervous System Diseases; Neurodegenerative Diseases; Brain Diseases | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine; Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Preladenant 1 mg BID (Experimental): Participants received preladenant 1 mg twice daily (BID) during the 12-week treatment period.
  Interventions: Drug: Preladenant; Drug: L-dopa; Drug: Other Parkinson's Disease treatments
- Preladenant 2 mg BID (Experimental): Participants received preladenant 2 mg BID during the 12-week treatment period.
  Interventions: Drug: Preladenant; Drug: L-dopa; Drug: Other Parkinson's Disease treatments
- Preladenant 5 mg BID (Experimental): Participants received preladenant 5 mg BID during the 12-week treatment period.
  Interventions: Drug: Preladenant; Drug: L-dopa; Drug: Other Parkinson's Disease treatments
- Preladenant 10 mg BID (Experimental): Participants received preladenant 10 mg BID during the 12-week treatment period.
  Interventions: Drug: Preladenant; Drug: L-dopa; Drug: Other Parkinson's Disease treatments
- Placebo BID (Placebo Comparator): Participants received preladenant matching placebo BID during the 12-week treatment period.
  Interventions: Drug: Placebo; Drug: L-dopa; Drug: Other Parkinson's Disease treatments

INTERVENTIONS:
Drug: Preladenant — 1 mg BID capsules
  Other Names: SCH 420814
  Arms: Preladenant 1 mg BID
Drug: Preladenant — 2 mg BID capsules
  Other Names: SCH 420814
  Arms: Preladenant 2 mg BID
Drug: Preladenant — 5 mg BID capsules
  Other Names: SCH 420814
  Arms: Preladenant 5 mg BID
Drug: Preladenant — 10 mg BID capsules
  Other Names: SCH 420814
  Arms: Preladenant 10 mg BID
Drug: Placebo — BID capsules
  Arms: Placebo BID
Drug: L-dopa — Participants must receive L-dopa as part of their usual ongoing treatment for Parkinson's Disease. L-dopa is often administered concomitantly with a dopa decarboxylase inhibitor (e.g., carbidopa).
Drug: Other Parkinson's Disease treatments — Participants may also receive other drugs as part of their usual ongoing treatment for Parkinson's Disease, such as dopamine agonists (e.g., pramipexole) and/or the catechol-O-methyl transferase (COMT) inhibitor entacapone.

SUMMARY:
The purpose of the study is to assess the efficacy and safety of a range of doses of SCH 420814 (preladenant) when used together with a stable dose of L-dopa/dopa decarboxylase inhibitor to treat Parkinson's disease. In this study, we will be comparing 3 doses (1 mg, 2 mg, and 5 mg taken twice a day) of preladenant with placebo (sugar pill). Following an Interim Analysis (temporary hold for new enrollment-ongoing subjects will continue on treatment) to review drug safety, a new dose group of 10 mg (taken twice a day) may be added.

Approximately 160 participants will be randomized in this study in approximately 22 study centers worldwide for the first part of this study. Following the Interim Analysis, 40 new participants may be added, for a total of 200 participants. The study is double blind, which means neither you nor your study doctor will know whether you are receiving the study medication or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 30 years of age, of either sex and of any race, with a diagnosis of moderate to severe idiopathic Parkinson's disease for at least 5 years.
* Women of childbearing potential must have a negative serum pregnancy test at Visit 2 (Week -1). If participant is postmenopausal (not surgically induced), she must be postmenopausal by history for at least 2 years before study entry. If not, proper birth control must be used.

Note: Acceptable methods of birth control include oral or injectable hormonal contraceptive, medically prescribed intrauterine device (IUD), and double-barrier method (eg, condom in combination with spermicide). Bilateral tubal ligation is an acceptable method of birth control for this study.

* Participants' clinical laboratory tests (complete blood count [CBC], blood chemistries, and urinalysis) must be within normal limits or clinically acceptable to the investigator/sponsor.

Exclusion Criteria:

* Participants with any form of drug-induced or atypical parkinsonism, cognitive impairment (Mini-Mental State Examination [MMSE] score <=23), a history of Diagnostic and Statistical Manual of Mental Disorders IV (DSM IV) diagnosed major depression, unstable mild depression or psychosis, or participants taking tolcapone will be excluded. (Participants with mild depression who are well controlled on a stable dose of an antidepressant medication for at least 4 weeks before screening will be eligible.)
* All participants with a severe or ongoing unstable medical condition will be excluded including those with a history of poorly controlled diabetes, obesity associated with metabolic syndrome, uncontrolled hypertension, cerebrovascular disease, or any form of clinically significant cardiac disease, symptomatic orthostatic hypotension, renal failure, history of abnormal renal function, seizures, alcohol/drug dependence, or previous surgery for Parkinson's disease.
* Average daily consumption of more than two 4-oz (120 mL) glasses of wine or their equivalent.
* Because it is not known whether preladenant passes into breast milk and because the effects, if any, of preladenant on the developing human are unknown, women who are breastfeeding or who are considering breastfeeding are excluded from this trial.
* Participants with allergy/sensitivity to study drug or its excipients.
* Participants with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study.
* Participants who have used any other investigational drugs within 30 days of Screening.
* Participants who are participating in any other clinical study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2006-11-20 (Actual); Primary Completion 2008-10-05 (Actual); Study Completion 2008-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Hauser RA, Cantillon M, Pourcher E, Micheli F, Mok V, Onofrj M, Huyck S, Wolski K. Preladenant in patients with Parkinson's disease and motor fluctuations: a phase 2, double-blind, randomised trial. Lancet Neurol. 2011 Mar;10(3):221-9. doi: 10.1016/S1474-4422(11)70012-6. PMID 21315654

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Started | 49 | 49 | 49 | 57 | 49
Treated | 49 | 49 | 47 | 54 | 47
Completed | 33 | 41 | 39 | 40 | 41
Not Completed | 16 | 8 | 10 | 17 | 8
Not completed — Adverse Event | 12 | 2 | 5 | 10 | 7
Not completed — Withdrawal by Subject | 3 | 4 | 2 | 2 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 2 | 0
Not completed — Did Not Meet Eligibility Criteria | 0 | 0 | 1 | 0 | 0
Not completed — Randomized in Error | 0 | 0 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of all participants who received at least one dose of study medication (either preladenant or placebo).
Groups:
- Preladenant 1 mg BID: Participants received preladenant 1 mg BID during the 12-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID | Total
Number analyzed (Participants) | 49 | 49 | 47 | 54 | 47 | 246
Age, Customized [Number; unit: Participants]
  Between 18 and 65 years | 30 | 25 | 24 | 32 | 27 | 138
  >=65 years | 19 | 24 | 23 | 22 | 20 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 17 | 22 | 16 | 87
  Male | 30 | 36 | 30 | 32 | 31 | 159

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint of 12 Weeks in the 3-day Average of Awake Time Per Day Spent in the "Off" State
Description: "Off" time refers to periods of inadequate control of Parkinson disease symptoms (worsening or presence of symptoms). For baseline and the 12 weeks treatment period, hours spent in the "off" state during awake time were recorded in half-hour time intervals using a daily diary at least 3 full days before scheduled visits. For baseline, the 24-hour average over 3 consecutive days was derived for Week -1. For endpoint, the 24-hour average was derived for the last available 3 consecutive days with postbaseline data available during the treatment period. Change from baseline in least squares (LS) means and pooled standard deviation (SD) were obtained from an analysis of covariance (ANCOVA) model with effect for treatment and baseline covariate. A negative change from baseline signifies less time spent in the "off" state.
Time Frame: Baseline (Week -1) and up to 12 weeks
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (awake time per day in the "off" state) was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
hours/day | -0.4 (2.48) | -1.3 (2.48) | -1.6 (2.48) | -1.7 (2.48) | -0.5 (2.48)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; LS means treatment difference in change from baseline to endpoint obtained from an ANCOVA model with effect for treatment and baseline covariate; Test type: Superiority or Other; p = 0.753, ANCOVA — The alpha threshold for statistical significance is 0.049 (2-sided); Difference in LS Means = 0.2, 95% CI 2-sided [-0.9 to 1.2]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; LS means treatment difference in change from baseline at endpoint obtained from an ANCOVA model with effect for treatment and baseline covariate; Test type: Superiority or Other; p = 0.162, ANCOVA — The alpha threshold for statistical significance is 0.049 (2-sided); Difference in LS Means = -0.7, 95% CI 2-sided [-1.7 to 0.3]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.049, ANCOVA — The alpha threshold for statistical significance is 0.049 (2-sided); Difference in LS Means = -1.0, 95% CI 2-sided [-2.1 to 0.0]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.019, ANCOVA — The alpha threshold for statistical significance is 0.049 (2-sided); Difference in LS Means = -1.2, 95% CI 2-sided [-2.2 to -0.2]

2. Secondary Outcome: Change From Baseline in Awake Time Per Day Spent in the "Off" State at Each Visit
Description: "Off" time refers to periods of inadequate control of Parkinson disease symptoms (worsening or presence of symptoms). Hours spent in the "off" state during awake time were recorded in half-hour time intervals using a daily diary at least 3 full days before scheduled visits. For baseline, the 24-hour average over 3 consecutive days was derived for Week -1. For treatment period visits, the 24-hour average was derived for the final 3 consecutive days with data available for the particular visit. Change from baseline in LS means and pooled SD were obtained from an ANCOVA model with treatment effect and baseline covariate. A negative change from baseline signifies less time spent in the "off" state.
Time Frame: Baseline (Week -1) and Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (awake time per day in the "off" state) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
hours/day
  Week 2 (n=46,47,43,49,45) | -0.3 (2.11) | -0.6 (2.11) | -1.0 (2.11) | -1.2 (2.11) | -0.2 (2.11)
  Week 4 (n=45,47,45,44,42) | -0.5 (2.36) | -1.1 (2.36) | -1.1 (2.36) | -0.9 (2.36) | -0.5 (2.36)
  Week 6 (n=39,46,42,41,42) | -0.3 (2.58) | -1.4 (2.58) | -1.3 (2.58) | -1.0 (2.58) | -0.8 (2.58)
  Week 8 (n=36,45,40,34,41) | -0.8 (2.34) | -1.2 (2.34) | -1.1 (2.34) | -1.7 (2.34) | -0.5 (2.34)
  Week 10 (n=35,42,40,36,41) | -0.3 (2.31) | -1.3 (2.31) | -1.7 (2.31) | -1.9 (2.31) | -0.4 (2.31)
  Week 12 (n=29,39,37,38,37) | -1.1 (2.42) | -1.4 (2.42) | -1.6 (2.42) | -1.9 (2.42) | -0.4 (2.42)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; LS means treatment difference in change from baseline to Week 2 obtained from an ANCOVA model with effect for treatment and baseline covariate; Test type: Superiority or Other; p = 0.935, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.9 to 0.8]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.326, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-1.3 to 0.4]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.070, ANCOVA; Difference in LS Means = -0.8, 95% CI 2-sided [-1.7 to 0.1]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.020, ANCOVA; Difference in LS Means = -1.0, 95% CI 2-sided [-1.9 to -0.2]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; LS means treatment difference in change from baseline to Week 4 obtained from an ANCOVA model with effect for treatment and baseline covariate; Test type: Superiority or Other; p = 0.982, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-1.0 to 1.0]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.281, ANCOVA; Difference in LS Means = -0.5, 95% CI 2-sided [-1.5 to 0.4]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.261, ANCOVA; Difference in LS Means = -0.6, 95% CI 2-sided [-1.6 to 0.4]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.447, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-1.4 to 0.6]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; LS means treatment difference in change from baseline to Week 6 obtained from an ANCOVA model with effect for treatment and baseline covariate; Test type: Superiority or Other; p = 0.378, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.6 to 1.6]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.299, ANCOVA; Difference in LS Means = -0.6, 95% CI 2-sided [-1.7 to 0.5]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.377, ANCOVA; Difference in LS Means = -0.5, 95% CI 2-sided [-1.6 to 0.6]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.707, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-1.3 to 0.9]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; LS means treatment difference in change from baseline to Week 8 obtained from an ANCOVA model with effect for treatment and baseline covariate; Test type: Superiority or Other; p = 0.562, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-1.4 to 0.7]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.156, ANCOVA; Difference in LS Means = -0.7, 95% CI 2-sided [-1.7 to 0.3]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.292, ANCOVA; Difference in LS Means = -0.5, 95% CI 2-sided [-1.6 to 0.5]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.034, ANCOVA; Difference in LS Means = -1.2, 95% CI 2-sided [-2.2 to -0.1]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; LS means treatment difference in change from baseline to Week 10 obtained from an ANCOVA model with effect for treatment and baseline covariate; Test type: Superiority or Other; p = 0.762, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-0.9 to 1.2]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.092, ANCOVA; Difference in LS Means = -0.9, 95% CI 2-sided [-1.9 to 0.1]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.013, ANCOVA; Difference in LS Means = -1.3, 95% CI 2-sided [-2.3 to -0.3]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.005, ANCOVA; Difference in LS Means = -1.5, 95% CI 2-sided [-2.5 to -0.4]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; LS means treatment difference in change from baseline to Week 12 obtained from an ANCOVA model with effect for treatment and baseline covariate; Test type: Superiority or Other; p = 0.293, ANCOVA; Difference in LS Means = -0.6, 95% CI 2-sided [-1.8 to 0.6]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.095, ANCOVA; Difference in LS Means = -0.9, 95% CI 2-sided [-2.0 to 0.2]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.040, ANCOVA; Difference in LS Means = -1.2, 95% CI [-2.3 to -0.1]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.011, ANCOVA; Difference in LS Means = -1.4, 95% CI 2-sided [-2.5 to -0.3]

3. Secondary Outcome: Change From Baseline in Awake Time Per Day Spent in the "on" State
Description: "On" time refers to periods of adequate control of Parkinson disease symptoms (symptoms better or absent). Hours spent in the "on" state during awake time were recorded in half-hour time intervals using a daily diary at least 3 full days before scheduled visits. For baseline, the 24-hour average over 3 consecutive days was derived for Week -1. For endpoint, the 24-hour average was derived for the last available 3 consecutive days with postbaseline data available during the treatment period. For treatment period visits, the 24-hour average was derived for the final 3 consecutive days with data available for the particular visit. Change from baseline in LS means and pooled SD were obtained from an ANCOVA model with effect for treatment and baseline covariate. A positive (+) change from baseline signifies more time spent in the "on" state.
Time Frame: Baseline (Week -1) and Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (awake time per day in the "on" state) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
hours/day
  Week 2 (n=46,47,43,49,45) | 0.4 (2.18) | 0.4 (2.18) | 0.9 (2.18) | 1.0 (2.18) | 0.1 (2.18)
  Week 4 (n=45,47,45,44,42) | 0.5 (2.45) | 0.6 (2.45) | 0.8 (2.45) | 0.7 (2.45) | 0.3 (2.45)
  Week 6 (n=39,46,42,41,42) | 0.3 (2.86) | 1.0 (2.86) | 1.0 (2.86) | 1.0 (2.86) | 0.6 (2.86)
  Week 8 (n=36,45,40,34,41) | 0.8 (2.59) | 1.0 (2.59) | 1.1 (2.59) | 1.1 (2.59) | 0.2 (2.59)
  Week 10 (n=35,42,40,34,41) | 0.2 (2.40) | 0.9 (2.40) | 1.5 (2.40) | 1.4 (2.40) | 0.1 (2.40)
  Week 12 (n=29,39,37,38,37) | 1.0 (2.64) | 0.8 (2.64) | 1.8 (2.64) | 1.4 (2.64) | 0.1 (2.64)
  Endpoint (n=47,48,45,49,45) | 0.4 (2.59) | 0.7 (2.59) | 1.4 (2.59) | 1.3 (2.59) | 0.2 (2.59)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.470, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.6 to 1.2]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.505, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.6 to 1.2]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.114, ANCOVA; Difference in LS Means = 0.7, 95% CI 2-sided [-0.2 to 1.7]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.042, ANCOVA; Difference in LS Means = 0.9, 95% CI 2-sided [0.0 to 1.8]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.684, ANCOVA; Difference in LS Means = 0.2, 94% CI 2-sided [-0.8 to 1.3]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.489, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.7 to 1.4]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.305, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.5 to 1.6]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.451, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.6 to 1.4]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.680, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-1.5 to 1.0]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.466, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.8 to 1.6]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.450, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.8 to 1.7]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.523, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.8 to 1.6]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.309, ANCOVA; Difference in LS Means = 0.6, 95% CI 2-sided [-0.6 to 1.8]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.136, ANCOVA; Difference in LS Means = 0.8, 95% CI 2-sided [-0.3 to 1.9]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.106, ANCOVA; Difference in LS Means = 0.9, 95% CI 2-sided [-0.2 to 2.1]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.144, ANCOVA; Difference in LS Means = 0.9, 95% CI 2-sided [-0.3 to 2.1]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.954, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.152, ANCOVA; Difference in LS Means = 0.8, 95% CI 2-sided [-0.3 to 1.8]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.012, ANCOVA; Difference in LS Means = 1.4, 95% CI 2-sided [0.3 to 2.4]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.025, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [0.2 to 2.3]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.151, ANCOVA; Difference in LS Means = 0.9, 95% CI 2-sided [-0.3 to 2.2]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.235, ANCOVA; Difference in LS Means = 0.7, 95% CI 2-sided [-0.5 to 1.9]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.007, ANCOVA; Difference in LS Means = 1.7, 95% CI 2-sided [0.5 to 2.9]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.033, ANCOVA; Difference in LS Means = 1.3, 95% CI 2-sided [0.1 to 2.5]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.757, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-0.9 to 1.2]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.341, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.5 to 1.6]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.024, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [0.2 to 2.3]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.049, ANCOVA; Difference in LS Means = 1.1, 95% CI 2-sided [0.0 to 2.1]

4. Secondary Outcome: Change From Baseline in Awake Time Per Day Spent in the "on" State (no Dyskinesias)
Description: "On" time refers to periods of adequate control of Parkinson disease symptoms (better/absent). Dyskinesias refers to maintenance therapy (e.g., L-dopa) side effects of chorea, dystonia, or in combination. Hours spent in the "on" state with no dyskinesias during awake time were recorded in half-hour time intervals using a daily diary at least 3 full days before scheduled visits. For baseline, the 24-hour average over 3 consecutive days was derived for Week -1. For endpoint, the 24-hour average was derived for the last available 3 consecutive days with postbaseline data available during the treatment period. For treatment period visits, the 24-hour average was derived for the final 3 consecutive days with data available for the particular visit. Change from baseline in LS means & pooled SD were obtained from an ANCOVA model with effect for treatment & baseline covariate. A (+) change from baseline signifies more time spent in the "on" state (no dyskinesias).
Time Frame: Baseline (Week -1) and Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (awake time per day in the "on" state with no dyskinesias) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
hours/day
  Week 2 (n=46,47,43,49,45) | 0.9 (2.54) | 0.1 (2.54) | 0.7 (2.54) | 0.3 (2.54) | 0.1 (2.54)
  Week 4 (n=45,47,45,44,42) | 0.8 (2.90) | 0.3 (2.90) | 0.6 (2.90) | 0.1 (2.90) | 0.1 (2.90)
  Week 6 (n=39,46,42,41,42) | 0.8 (3.31) | 0.4 (3.31) | 0.9 (3.31) | 0.2 (3.31) | 0.3 (3.31)
  Week 8 (n=36,45,40,34,41) | 1.1 (3.28) | 0.0 (3.28) | 1.0 (3.28) | 0.1 (3.28) | 0.5 (3.28)
  Week 10 (n=35,42,40,36,41) | 0.7 (3.40) | 0.1 (3.40) | 1.4 (3.40) | 0.6 (3.40) | 0.6 (3.40)
  Week 12 (n=29,39,37,38,37) | 1.2 (3.70) | 0.2 (3.70) | 1.4 (3.70) | 0.5 (3.70) | 0.9 (3.70)
  Endpoint (n=47,48,45,49,45) | 1.0 (3.58) | 0.2 (3.58) | 1.2 (3.58) | 0.7 (3.58) | 0.9 (3.58)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.151, ANCOVA; Difference in LS Means = 0.8, 95% CI 2-sided [-0.3 to 1.8]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.930, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-1.1 to 1.0]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.343, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.6 to 1.6]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.746, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-0.9 to 1.2]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.222, ANCOVA; Difference in LS Means = 0.8, 94% CI 2-sided [-0.5 to 2.0]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.673, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-1.0 to 1.5]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.415, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.7 to 1.7]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.968, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-1.3 to 1.2]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.543, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-1.0 to 1.9]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.967, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-1.4 to 1.4]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.411, ANCOVA; Difference in LS Means = 0.6, 95% CI 2-sided [-0.8 to 2.0]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.864, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-1.6 to 1.3]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.449, ANCOVA; Difference in LS Means = 0.6, 95% CI 2-sided [-0.9 to 2.0]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.411, ANCOVA; Difference in LS Means = -0.6, 95% CI 2-sided [-2.0 to 0.8]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.576, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-1.0 to 1.8]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.603, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-1.9 to 1.1]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.842, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-1.4 to 1.7]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.558, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-1.9 to 1.0]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.245, ANCOVA; Difference in LS Means = 0.9, 95% CI 2-sided [-0.6 to 2.4]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.930, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-1.5 to 1.6]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.759, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-1.5 to 2.1]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.374, ANCOVA; Difference in LS Means = -0.8, 95% CI 2-sided [-2.4 to 0.9]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.621, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-1.3 to 2.1]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.607, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-2.1 to 1.2]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.907, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-1.4 to 1.6]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.368, ANCOVA; Difference in LS Means = -0.7, 95% CI 2-sided [-2.1 to 0.8]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.654, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-1.1 to 1.8]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.769, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-1.7 to 1.2]

5. Secondary Outcome: Change From Baseline in Awake Time Per Day Spent in the "on" State (With Troublesome Dyskinesias)
Description: "On" time refers to periods of adequate control of Parkinson disease symptoms (better/absent). Troublesome dyskinesias refers to maintenance therapy side effects of chorea, dystonia, or in combination that impair function. Hours spent in the "on" state with troublesome dyskinesias during awake time were recorded in half-hour time intervals using a daily diary at least 3 full days before scheduled visits. For baseline, the 24-hour average over 3 consecutive days was derived for Week -1. For endpoint, the 24-hour average was derived for the last available 3 consecutive days with postbaseline data available during the treatment period. For treatment period visits, the 24-hour average was derived for the final 3 consecutive days with data available for the particular visit. Change from baseline in LS means & pooled SD were obtained using ANCOVA with treatment effect & baseline covariate. A (+) change from baseline signifies more time spent in the "on" state (troublesome dyskinesias).
Time Frame: Baseline (Week -1) and Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (awake time per day in the "on" state with troublesome dyskinesias) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
hours/day
  Week 2 (n=46,47,43,49,45) | -0.2 (1.21) | -0.2 (1.21) | 0.0 (1.21) | 0.2 (1.21) | 0.3 (1.21)
  Week 4 (n=45,47,45,44,42) | -0.1 (1.39) | 0.0 (1.39) | 0.0 (1.39) | 0.2 (1.39) | 0.2 (1.39)
  Week 6 (n=39,46,42,41,42) | -0.2 (1.81) | 0.1 (1.81) | -0.3 (1.81) | 0.2 (1.81) | 0.3 (1.81)
  Week 8 (n=36,45,40,34,41) | -0.2 (1.65) | 0.2 (1.65) | 0.0 (1.65) | 0.1 (1.65) | 0.1 (1.65)
  Week 10 (n=35,42,40,36,41) | -0.3 (1.61) | 0.1 (1.61) | -0.1 (1.61) | 0.1 (1.61) | 0.1 (1.61)
  Week 12 (n=29,39,37,38,37) | 0.0 (1.84) | 0.2 (1.84) | 0.2 (1.84) | 0.4 (1.84) | 0.1 (1.84)
  Endpoint (n=47,48,45,49,45) | -0.1 (1.79) | 0.1 (1.79) | 0.1 (1.79) | 0.4 (1.79) | 0.1 (1.79)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.055, ANCOVA; Difference in LS Means = -0.5, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.071, ANCOVA; Difference in LS Means = -0.5, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.288, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-0.8 to 0.2]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.764, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-0.6 to 0.4]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.342, ANCOVA; Difference in LS Means = -0.3, 94% CI 2-sided [-0.9 to 0.3]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.611, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-0.7 to 0.4]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.424, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.991, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.6 to 0.6]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.185, ANCOVA; Difference in LS Means = -0.5, 95% CI 2-sided [-1.3 to 0.3]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.597, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-1.0 to 0.6]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.090, ANCOVA; Difference in LS Means = -0.7, 95% CI 2-sided [-1.5 to 0.1]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.686, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-0.9 to 0.6]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.501, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-1.0 to 0.5]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.764, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.6 to 0.8]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.715, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-0.9 to 0.6]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.924, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.7 to 0.8]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.264, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-1.2 to 0.3]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.976, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.7 to 0.7]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.626, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-0.9 to 0.5]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.925, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.8 to 0.7]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.849, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-1.0 to 0.8]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.755, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.7 to 1.0]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.863, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.8 to 0.9]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.477, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.5 to 1.1]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.432, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-1.0 to 0.4]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.909, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.8 to 0.7]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.812, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-0.8 to 0.7]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.540, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-0.5 to 1.0]

6. Secondary Outcome: Change From Baseline in Awake Time Per Day Spent in the "on" State (Without Troublesome Dyskinesias)
Description: "On" time refers to periods of adequate control of Parkinson disease symptoms (better/absent). Troublesome dyskinesias refers to maint. therapy side effects of chorea, dystonia, or in combination that impair function. Hours spent in the "on" state without troubles. dyskinesias during awake time were recorded in half-hour time intervals using a daily diary at least 3 full days before scheduled visits. For baseline, the 24-hour average over 3 consecutive days was derived for Week -1. For endpoint, the 24-hour average was derived for the last available 3 consecutive days with postbaseline data available during the treatment period. For treatment period visits, the 24-hour average was derived for the final 3 consecutive days with data available for the particular visit. Change from baseline in LS means & pooled SD were obtained using ANCOVA with treatment effect & baseline covariate. A (+) change from baseline signifies more time spent in the "on" state (without troubles. dyskinesias).
Time Frame: Baseline (Week -1) and Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (awake time per day in the "on" state without troublesome dyskinesias) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
hours/day
  Week 2 (n=46,47,43,49,45) | -0.3 (1.95) | 0.5 (1.95) | 0.2 (1.95) | 0.5 (1.95) | -0.3 (1.95)
  Week 4 (n=45,47,45,44,42) | -0.2 (2.31) | 0.2 (2.31) | 0.3 (2.31) | 0.4 (2.31) | 0.0 (2.31)
  Week 6 (n=39,46,42,41,42) | -0.2 (2.64) | 0.5 (2.64) | 0.5 (2.64) | 0.5 (2.64) | -0.1 (2.64)
  Week 8 (n=36,45,40,34,41) | -0.1 (2.73) | 0.8 (2.73) | 0.3 (2.73) | 0.8 (2.73) | -0.5 (2.73)
  Week 10 (n=35,42,40,36,41) | -0.2 (2.64) | 0.7 (2.64) | 0.2 (2.64) | 0.7 (2.64) | -0.5 (2.64)
  Week 12 (n=29,39,37,38,37) | -0.2 (2.73) | 0.4 (2.73) | 0.2 (2.73) | 0.5 (2.73) | -1.0 (2.73)
  Endpoint (n=47,48,45,49,45 | -0.4 (2.59) | 0.4 (2.59) | 0.2 (2.59) | 0.2 (2.59) | -0.8 (2.59)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.829, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.7 to 0.9]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.042, ANCOVA; Difference in LS Means = 0.8, 95% CI 2-sided [0.0 to 1.6]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.204, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.3 to 1.4]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.035, ANCOVA; Difference in LS Means = 0.9, 95% CI 2-sided [0.1 to 1.6]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.696, ANCOVA; Difference in LS Means = -0.2, 94% CI 2-sided [-1.2 to 0.8]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.625, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-0.7 to 1.2]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.478, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.6 to 1.3]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.380, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.5 to 1.4]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.925, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-1.2 to 1.1]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.285, ANCOVA; Difference in LS Means = 0.6, 95% CI 2-sided [-0.5 to 1.7]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.296, ANCOVA; Difference in LS Means = 0.6, 95% CI 2-sided [-0.5 to 1.7]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.241, ANCOVA; Difference in LS Means = 0.7, 95% CI 2-sided [-0.5 to 1.8]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.571, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.9 to 1.6]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.032, ANCOVA; Difference in LS Means = 1.3, 95% CI 2-sided [0.1 to 2.4]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.214, ANCOVA; Difference in LS Means = 0.8, 95% CI 2-sided [-0.4 to 2.0]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.051, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [0.0 to 2.5]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.572, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.9 to 1.5]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.041, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [0.1 to 2.4]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.240, ANCOVA; Difference in LS Means = 0.7, 95% CI 2-sided [-0.5 to 1.9]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.047, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [0.0 to 2.4]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.228, ANCOVA; Difference in LS Means = 0.8, 95% CI 2-sided [-0.5 to 2.2]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.030, ANCOVA; Difference in LS Means = 1.4, 95% CI 2-sided [0.1 to 2.6]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.059, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [0.0 to 2.5]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.021, ANCOVA; Difference in LS Means = 1.5, 95% CI 2-sided [0.2 to 2.7]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.428, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.6 to 1.5]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.025, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [0.2 to 2.3]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.064, ANCOVA; Difference in LS Means = 1.0, 95% CI 2-sided [-0.1 to 2.1]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.047, ANCOVA; Difference in LS Means = 1.1, 95% CI 2-sided [0.0 to 2.1]

7. Secondary Outcome: Change From Baseline in Absolute Duration of Dyskinesias
Description: Dyskinesias refers to maintenance therapy side effects of chorea, dystonia, or in combination (that occur in the ON time). Hours spent with dyskinesias (troublesome and not troublesome) were recorded in half-hour time intervals using a daily diary at least 3 full days before scheduled visits. For baseline, the 24-hour average over 3 consecutive days was derived for Week -1. For endpoint, the 24-hour average was derived for the last available 3 consecutive days with postbaseline data available during the treatment period. For treatment period visits, the 24-hour average was derived for the final 3 consecutive days with data available for the particular visit. Change from baseline in LS means & pooled SD were obtained using ANCOVA with treatment effect & baseline covariate. A negative change from baseline signifies less time spent with dyskinesia.
Time Frame: Baseline (Week -1) and Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (awake time per day in the "on" state with troublesome and not troblesome dyskinesias) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
hours/day
  Week 2 (n=46,47,43,49,45) | -0.5 (2.26) | 0.3 (2.26) | 0.2 (2.26) | 0.7 (2.26) | 0.0 (2.26)
  Week 4 (n=45,47,45,44,42) | -0.4 (2.81) | 0.2 (2.81) | 0.3 (2.81) | 0.6 (2.81) | 0.2 (2.81)
  Week 6 (n=39,46,42,41,42) | -0.5 (3.25) | 0.6 (3.25) | 0.2 (3.25) | 0.7 (3.25) | 0.2 (3.25)
  Week 8 (n=36,45,40,34,41) | -0.3 (3.25) | 1.0 (3.25) | 0.2 (3.25) | 0.9 (3.25) | -0.3 (3.25)
  Week 10 (n=35,42,40,36,41) | -0.5 (3.11) | 0.8 (3.11) | 0.1 (3.11) | 0.8 (3.11) | -0.4 (3.11)
  Week 12 (n=29,39,37,38,37) | -0.2 (3.27) | 0.6 (3.27) | 0.4 (3.27) | 0.9 (3.27) | -0.9 (3.27)
  Endpoint (n=47,48,45,49,45 | -0.6 (3.18) | 0.5 (3.18) | 0.2 (3.18) | 0.6 (3.18) | -0.7 (3.18)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.345, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-1.4 to 0.5]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.468, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.6 to 1.3]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.596, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.7 to 1.2]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.107, ANCOVA; Difference in LS Means = 0.8, 95% CI 2-sided [-0.2 to 1.7]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.348, ANCOVA; Difference in LS Means = -0.6, 94% CI 2-sided [-1.8 to 0.6]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.938, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-1.1 to 1.2]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.897, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-1.1 to 1.3]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.518, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.8 to 1.6]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.311, ANCOVA; Difference in LS Means = -0.7, 95% CI 2-sided [-2.2 to 0.7]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.597, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-1.0 to 1.7]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.925, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-1.5 to 1.3]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.478, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.9 to 1.9]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.995, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-1.5 to 1.5]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.057, ANCOVA; Difference in LS Means = 1.3, 95% CI 2-sided [0.0 to 2.7]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.431, ANCOVA; Difference in LS Means = 0.6, 95% CI 2-sided [-0.9 to 2.0]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.099, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [-0.2 to 2.7]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.847, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-1.5 to 1.3]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.093, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [-0.2 to 2.5]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.471, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.9 to 1.9]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.102, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [-0.2 to 2.6]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.415, ANCOVA; Difference in LS Means = 0.7, 95% CI 2-sided [-0.9 to 2.3]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.051, ANCOVA; Difference in LS Means = 1.5, 95% CI 2-sided [0.0 to 3.0]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.103, ANCOVA; Difference in LS Means = 1.3, 95% CI 2-sided [-0.3 to 2.8]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.022, ANCOVA; Difference in LS Means = 1.7, 95% CI 2-sided [0.3 to 3.2]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.903, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-1.2 to 1.4]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.074, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [-0.1 to 2.5]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.185, ANCOVA; Difference in LS Means = 0.9, 95% CI 2-sided [-0.4 to 2.2]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.054, ANCOVA; Difference in LS Means = 1.3, 95% CI 2-sided [0.0 to 2.6]

8. Secondary Outcome: Change From Baseline in Total Sleep Time
Description: Hours spent in the sleep state were recorded using a daily diary at least 3 full days before scheduled visit. For baseline, the 24-hour average over 3 consecutive days was derived for Week -1. For endpoint, the 24-hour average was derived for the last available 3 consecutive days with postbaseline data available during the treatment period. For treatment period visits, the 24-hour average was derived for the final 3 consecutive days with data available for the particular visit. Change from baseline in LS means & pooled SD were obtained using ANCOVA with treatment effect & baseline covariate. A positive change from baseline means more time asleep and a negative change means less time asleep.
Time Frame: Baseline (Week -1) and Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (total sleep time) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
hours/day
  Week 2 (n=46,47,43,49,45) | 0.0 (1.14) | 0.2 (1.14) | 0.1 (1.14) | 0.1 (1.14) | 0.0 (1.14)
  Week 4 (n=45,47,45,44,42) | 0.1 (1.23) | 0.5 (1.23) | 0.1 (1.23) | 0.2 (1.23) | 0.1 (1.23)
  Week 6 (n=39,46,42,41,42) | 0.1 (1.28) | 0.4 (1.28) | -0.1 (1.28) | 0.1 (1.28) | 0.2 (1.28)
  Week 8 (n=36,45,40,34,41) | 0.1 (1.43) | 0.2 (1.43) | 0.1 (1.43) | 0.2 (1.43) | 0.2 (1.43)
  Week 10 (n=35,42,40,36,41) | 0.2 (1.34) | 0.3 (1.34) | 0.3 (1.34) | 0.5 (1.34) | 0.2 (1.34)
  Week 12 (n=29,39,37,38,37) | 0.2 (1.24) | 0.5 (1.24) | 0.0 (1.24) | 0.3 (1.24) | 0.2 (1.24)
  Endpoint (n=47,48,45,49,45) | 0.2 (1.33) | 0.5 (1.33) | 0.1 (1.33) | 0.2 (1.33) | 0.1 (1.33)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.985, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.5 to 0.5]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.556, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.3 to 0.6]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.776, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.777, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.920, ANCOVA; Difference in LS Means = 0.0, 94% CI 2-sided [-0.5 to 0.5]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.155, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.843, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.673, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.612, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-0.7 to 0.4]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.512, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-0.4 to 0.7]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.269, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-0.9 to 0.2]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.516, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-0.7 to 0.4]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.597, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-0.8 to 0.5]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.766, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-0.7 to 0.5]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.428, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-0.9 to 0.4]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.796, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.988, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.6 to 0.6]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.786, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.702, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.371, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.3 to 0.9]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.981, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.6 to 0.6]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.282, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.3 to 0.9]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.550, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-0.7 to 0.4]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.720, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.742, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.211, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.2 to 0.9]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.906, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.6 to 0.5]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.868, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.5 to 0.6]

9. Secondary Outcome: Change From Baseline in Frequency of Sleep Attacks at Week 2
Description: Sleep attacks are uncontrollable episodes of sleep that occur during the daytime lasting a few seconds to several minutes. A questionnaire to determine sleep attacks over the prior 2 week period was administered at baseline and at 2-week intervals during the treatment period. Frequency of sleep attacks over the two-week treatment period intervals were tabulated in relation to the baseline assessment. Results are presented as participants showing the respective change in frequency of sleep attacks at baseline to the week of assessment (Week 2) (as reported by the participant). For example, someone who had >2 sleep attacks at BL who had a decrease of 1-2 by Week 2 would be reported as BL >2 to WK2 1-2. BL = baseline. WK = week.
Time Frame: Baseline (predose Day 1) and 2 hours postdose at Week 2
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (sleep attacks) for the assessment week was used for analysis.
Measure: Number; unit: Participants
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
Participants
  BL 0 to WK2 <-2 (n=36,42,39,43,41) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK2 -1,-2 (n=36,42,39,43,41) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK2 0 (n=36,42,39,43,41) | 31 | 39 | 36 | 41 | 37
  BL 0 to WK2 1,2 (n=36,42,39,43,41) | 3 | 1 | 1 | 1 | 1
  BL 0 to WK2 >-2 (n=36,42,39,43,41) | 2 | 2 | 2 | 1 | 3
  BL 1,2 to WK2 <-2 (n=4,2,2,2,1) | 0 | 0 | 1 | 0 | 0
  BL 1,2 to WK2 -1,-2 (n=4,2,2,2,1) | 2 | 1 | 1 | 0 | 0
  BL 1,2 to WK2 0 (n=4,2,2,2,1) | 1 | 1 | 0 | 0 | 1
  BL 1,2 to WK2 1,2 (n=4,2,2,2,1) | 0 | 0 | 0 | 1 | 0
  BL 1,2 to WK2 >-2 (n=4,2,2,2,1) | 1 | 0 | 0 | 1 | 0
  BL >2 to WK2 <-2 (n=6,2,4,0,2) | 3 | 0 | 2 | 0 | 1
  BL >2 to WK2 -1,-2 (n=6,2,4,0,2) | 0 | 1 | 0 | 0 | 0
  BL >2 to WK2 0 (n=6,2,4,0,2) | 3 | 0 | 1 | 0 | 0
  BL >2 to WK2 1,2 (n=6,2,4,0,2) | 0 | 1 | 0 | 0 | 0
  BL >2 to WK2 >-2 (n=6,2,4,0,2) | 0 | 0 | 1 | 0 | 1

10. Secondary Outcome: Change From Baseline in Frequency of Sleep Attacks at Week 4
Description: Sleep attacks are uncontrollable episodes of sleep that occur during the daytime lasting a few seconds to several minutes. A questionnaire to determine sleep attacks over the prior 2 week period was administered at baseline and at 2-week intervals during the treatment period. Frequency of sleep attacks over the two-week treatment period intervals were tabulated in relation to the baseline assessment. Results are presented as participants showing the respective change in frequency of sleep attacks at baseline to the week of assessment (Week 4) (as reported by the participant). For example, someone who had >2 sleep attacks at BL who had a decrease of 1-2 by Week 4 would be reported as BL >2 to WK4 1-2. BL = baseline. WK = week.
Time Frame: Baseline (predose Day 1) and 2 hours postdose at Week 4
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
Participants
  BL 0 to WK4 <-2 (n=32,43,39,43,39) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK4 -1,-2 (n=32,43,39,43,39) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK4 0 (n=32,43,39,43,39) | 30 | 40 | 34 | 40 | 36
  BL 0 to WK4 1,2 (n=32,43,39,43,39) | 1 | 3 | 3 | 2 | 1
  BL 0 to WK4 >-2 (n=32,43,39,43,39) | 1 | 0 | 2 | 1 | 2
  BL 1,2 to WK4 <-2 (n=3,2,2,1,1) | 1 | 0 | 1 | 0 | 1
  BL 1,2 to WK4 -1,-2 (n=3,2,2,1,1) | 1 | 0 | 0 | 1 | 0
  BL 1,2 to WK4 0 (n=3,2,2,1,1) | 0 | 1 | 1 | 0 | 0
  BL 1,2 to WK4 1,2 (n=3,2,2,1,1) | 1 | 1 | 0 | 0 | 0
  BL 1,2 to WK4 >-2 (n=3,2,2,1,1) | 0 | 0 | 0 | 0 | 0
  BL >2 to WK4 <-2 (n=6,2,4,0,2) | 5 | 1 | 2 | 0 | 1
  BL >2 to WK4 -1,-2 (n=6,2,4,0,2) | 0 | 1 | 0 | 0 | 0
  BL >2 to WK4 0 (n=6,2,4,0,2) | 0 | 0 | 0 | 0 | 1
  BL >2 to WK4 1,2 (n=6,2,4,0,2) | 1 | 0 | 1 | 0 | 0
  BL >2 to WK4 >-2 (n=6,2,4,0,2) | 0 | 0 | 1 | 0 | 0

11. Secondary Outcome: Change From Baseline in Frequency of Sleep Attacks at Week 6
Description: Sleep attacks are uncontrollable episodes of sleep that occur during the daytime lasting a few seconds to several minutes. A questionnaire to determine sleep attacks over the prior 2 week period was administered at baseline and at 2-week intervals during the treatment period. Frequency of sleep attacks over the two-week treatment period intervals were tabulated in relation to the baseline assessment. Results are presented as participants showing the respective change in frequency of sleep attacks at baseline to the week of assessment (Week 6) (as reported by the participant). For example, someone who had >2 sleep attacks at BL who had a decrease of 1-2 by Week 6 would be reported as BL >2 to WK6 1-2. BL = baseline. WK = week.
Time Frame: Baseline (predose Day 1) and 2 hours postdose at Week 6
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
Participants
  BL 0 to WK6 <-2 (n=30,39,37,34,39) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK6 -1,-2 (n=30,39,37,34,39) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK6 0 (n=30,39,37,34,39) | 28 | 38 | 32 | 34 | 36
  BL 0 to WK6 1,2 (n=30,39,37,34,39) | 1 | 0 | 1 | 0 | 2
  BL 0 to WK6 >-2 (n=30,39,37,34,39) | 1 | 1 | 4 | 0 | 1
  BL 1,2 to WK6 <-2 (n=4,2,2,1,1) | 1 | 1 | 2 | 0 | 1
  BL 1,2 to WK6 -1,-2 (n=4,2,2,1,1) | 1 | 0 | 0 | 1 | 0
  BL 1,2 to WK6 0 (n=4,2,2,1,1) | 0 | 1 | 0 | 0 | 0
  BL 1,2 to WK6 1,2 (n=4,2,2,1,1) | 1 | 0 | 0 | 0 | 0
  BL 1,2 to WK6 >-2 (n=4,2,2,1,1) | 1 | 0 | 0 | 0 | 0
  BL >2 to WK6 <-2 (n=6,2,4,0,2) | 5 | 1 | 3 | 0 | 1
  BL >2 to WK6 -1,-2 (n=6,2,4,0,2) | 0 | 1 | 0 | 0 | 0
  BL >2 to WK6 0 (n=6,2,4,0,2) | 0 | 0 | 0 | 0 | 0
  BL >2 to WK6 1,2 (n=6,2,4,0,2) | 1 | 0 | 0 | 0 | 0
  BL >2 to WK6 >-2 (n=6,2,4,0,2) | 0 | 0 | 1 | 0 | 1

12. Secondary Outcome: Change From Baseline in Frequency of Sleep Attacks at Week 8
Description: Sleep attacks are uncontrollable episodes of sleep that occur during the daytime lasting a few seconds to several minutes. A questionnaire to determine sleep attacks over the prior 2 week period was administered at baseline and at 2-week intervals during the treatment period. Frequency of sleep attacks over the two-week treatment period intervals were tabulated in relation to the baseline assessment. Results are presented as participants showing the respective change in frequency of sleep attacks at baseline to the week of assessment (Week 8) (as reported by the participant). For example, someone who had >2 sleep attacks at BL who had a decrease of 1-2 by Week 8 would be reported as BL >2 to WK8 1-2. BL = baseline. WK = week.
Time Frame: Baseline (predose Day 1) and 2 hours postdose at Week 8
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
Participants
  BL 0 to WK8 <-2 (n=27,39,35,37,39) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK8 -1,-2 (n=27,39,35,37,39) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK8 0 (n=27,39,35,37,39) | 24 | 37 | 33 | 36 | 36
  BL 0 to WK8 1,2 (n=27,39,35,37,39) | 2 | 2 | 1 | 0 | 1
  BL 0 to WK8 >-2 (n=27,39,35,37,39) | 1 | 0 | 1 | 1 | 2
  BL 1,2 to WK8 <-2 (n=2,2,2,1,0) | 0 | 1 | 2 | 0 | 0
  BL 1,2 to WK8 -1,-2 (n=2,2,2,1,0) | 1 | 0 | 0 | 0 | 0
  BL 1,2 to WK8 0 (n=2,2,2,1,0) | 1 | 0 | 0 | 0 | 0
  BL 1,2 to WK8 1,2 (n=2,2,2,1,0) | 0 | 1 | 0 | 1 | 0
  BL 1,2 to WK8 >-2 (n=2,2,2,1,0) | 0 | 0 | 0 | 0 | 0
  BL >2 to WK8 <-2 (n=5,2,4,0,2) | 3 | 2 | 4 | 0 | 1
  BL >2 to WK8 -1,-2 (n=5,2,4,0,2) | 0 | 0 | 0 | 0 | 0
  BL >2 to WK8 0 (n=5,2,4,0,2) | 1 | 0 | 0 | 0 | 0
  BL >2 to WK8 1,2 (n=5,2,4,0,2) | 1 | 0 | 0 | 0 | 0
  BL >2 to WK8 >-2 (n=5,2,4,0,2) | 0 | 0 | 0 | 0 | 1

13. Secondary Outcome: Change From Baseline in Frequency of Sleep Attacks at Week 10
Description: Sleep attacks are uncontrollable episodes of sleep that occur during the daytime lasting a few seconds to several minutes. A questionnaire to determine sleep attacks over the prior 2 week period was administered at baseline and at 2-week intervals during the treatment period. Frequency of sleep attacks over the two-week treatment period intervals were tabulated in relation to the baseline assessment. Results are presented as participants showing the respective change in frequency of sleep attacks at baseline to the week of assessment (Week 10) (as reported by the participant). For example, someone who had >2 sleep attacks at BL who had a decrease of 1-2 by Week 10 would be reported as BL >2 to WK10 1-2. BL = baseline. WK = week.
Time Frame: Baseline (predose Day 1) and 2 hours postdose at Week 10
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
Participants
  BL 0 to WK10 <-2 (n=25,36,34,35,38) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK10 -1,-2 (n=25,36,34,35,38) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK10 0 (n=25,36,34,35,38) | 21 | 35 | 31 | 35 | 36
  BL 0 to WK10 1,2 (n=25,36,34,35,38) | 4 | 1 | 3 | 0 | 0
  BL 0 to WK10 >-2 (n=25,36,34,35,38) | 0 | 0 | 0 | 0 | 2
  BL 1,2 to WK10 <-2 (n=3,2,2,1,1) | 0 | 1 | 2 | 0 | 0
  BL 1,2 to WK10 -1,-2 (n=3,2,2,1,1) | 1 | 1 | 0 | 1 | 1
  BL 1,2 to WK10 0 (n=3,2,2,1,1) | 1 | 0 | 0 | 0 | 0
  BL 1,2 to WK10 1,2 (n=3,2,2,1,1) | 1 | 0 | 0 | 0 | 0
  BL 1,2 to WK10 >-2 (n=3,2,2,1,1) | 0 | 0 | 0 | 0 | 0
  BL >2 to WK10 <-2 (n=5,2,4,0,2) | 4 | 2 | 3 | 0 | 1
  BL >2 to WK10 -1,-2 (n=5,2,4,0,2) | 0 | 0 | 0 | 0 | 0
  BL >2 to WK10 0 (n=5,2,4,0,2) | 1 | 0 | 0 | 0 | 0
  BL >2 to WK10 1,2 (n=5,2,4,0,2) | 0 | 0 | 1 | 0 | 0
  BL >2 to WK10 >-2 (n=5,2,4,0,2) | 0 | 0 | 0 | 0 | 1

14. Secondary Outcome: Change From Baseline in Frequency of Sleep Attacks at Week 12
Description: Sleep attacks are uncontrollable episodes of sleep that occur during the daytime lasting a few seconds to several minutes. A questionnaire to determine sleep attacks over the prior 2 week period was administered at baseline and at 2-week intervals during the treatment period. Frequency of sleep attacks over the two-week treatment period intervals were tabulated in relation to the baseline assessment. Results are presented as participants showing the respective change in frequency of sleep attacks at baseline to the week of assessment (Week 12) (as reported by the participant). For example, someone who had >2 sleep attacks at BL who had a decrease of 1-2 by Week 12 would be reported as BL >2 to WK12 1-2. BL = baseline. WK = week.
Time Frame: Baseline (predose Day 1) and 2 hours postdose at Week 12
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
Participants
  BL 0 to WK12 <-2 (n=24,36,33,39,37) | 0 | 0 | 0 | 1 | 0
  BL 0 to WK12 -1,-2 (n=24,36,33,39,37) | 0 | 0 | 0 | 0 | 0
  BL 0 to WK12 0 (n=24,36,33,39,37) | 21 | 35 | 31 | 35 | 34
  BL 0 to WK12 1,2 (n=24,36,33,39,37) | 2 | 1 | 0 | 3 | 1
  BL 0 to WK12 >-2 (n=24,36,33,39,37) | 1 | 0 | 2 | 0 | 2
  BL 1,2 to WK12 <-2 (n=3,2,2,1,1) | 0 | 0 | 2 | 0 | 1
  BL 1,2 to WK12 -1,-2 (n=3,2,2,1,1) | 2 | 0 | 0 | 0 | 0
  BL 1,2 to WK12 0 (n=3,2,2,1,1) | 0 | 1 | 0 | 0 | 0
  BL 1,2 to WK12 1,2 (n=3,2,2,1,1) | 1 | 1 | 0 | 1 | 0
  BL 1,2 to WK12 >-2 (n=3,2,2,1,1) | 0 | 0 | 0 | 0 | 0
  BL >2 to WK12 <-2 (n=4,2,4,0,2) | 2 | 1 | 3 | 0 | 1
  BL >2 to WK12 -1,-2 (n=4,2,4,0,2) | 0 | 1 | 0 | 0 | 0
  BL >2 to WK12 0 (n=4,2,4,0,2) | 1 | 0 | 0 | 0 | 0
  BL >2 to WK12 1,2 (n=4,2,4,0,2) | 1 | 0 | 1 | 0 | 1
  BL >2 to WK12 >-2 (n=4,2,4,0,2) | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part 1
Description: The UPDRS is a frequently used multi-item 4-part questionnaire designed to assess various aspects of Parkinson's disease severity. A total of 42 items are assessed divided across Parts 1 to 4. Part 1 assesses mentation (4 items scored from 0 [best] to 4 [worst]; total range 0-16). Assessments were obtained at baseline (predose Day 1) and 2 hours postdose at Weeks 2, 4, 6, 8, 10, and 12. For endpoint, the last postbaseline visit while on study medication was used. Change from baseline in LS means and pooled SD were obtained from an ANCOVA model with effect for treatment and baseline covariate. Negative change from baseline indicates a decrease in severity.
Time Frame: Baseline (predose Day 1) and 2 hours postdose at Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (UPDRS Part 1) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
Units on a Scale
  Week 2 (n=44,42,40,41,41) | 0.1 (1.18) | -0.2 (1.18) | -0.2 (1.18) | -0.5 (1.18) | 0.2 (1.18)
  Week 4 (n=40,45,41,43,43) | -0.1 (1.24) | 0.0 (1.24) | -0.2 (1.24) | -0.2 (1.24) | 0.2 (1.24)
  Week 6 (n=39,41,39,35,42) | -0.1 (1.16) | -0.1 (1.16) | -0.4 (1.16) | -0.2 (1.16) | 0.3 (1.16)
  Week 8 (n=33,42,38,37,41) | 0.2 (1.21) | -0.1 (1.21) | -0.5 (1.21) | -0.2 (1.21) | 0.1 (1.21)
  Week 10 (n=32,39,37,35,41) | 0.2 (1.19) | 0.1 (1.19) | -0.5 (1.19) | 0.0 (1.19) | -0.1 (1.19)
  Week 12 (n=31,37,36,38,37) | 0.0 (1.23) | -0.1 (1.23) | -0.6 (1.23) | -0.3 (1.23) | 0.2 (1.23)
  Endpoint (n=45,46,41,47,44) | 0.1 (1.28) | 0.1 (1.28) | -0.5 (1.28) | -0.2 (1.28) | 0.3 (1.28)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.747, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-0.6 to 0.4]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.140, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-0.9 to 0.1]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.148, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-0.9 to 0.1]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.005, ANCOVA; Difference in LS Means = -0.7, 95% CI 2-sided [-1.2 to -0.2]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.256, ANCOVA; Difference in LS Means = -0.3, 94% CI 2-sided [-0.8 to 0.2]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.343, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.102, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-1.0 to 0.1]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.161, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-0.9 to 0.2]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.150, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-0.9 to 0.1]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.175, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-0.9 to 0.2]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.013, ANCOVA; Difference in LS Means = -0.7, 95% CI 2-sided [-1.2 to -0.1]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.120, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-0.9 to 0.1]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.971, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.6 to 0.6]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.456, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-0.7 to 0.3]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.018, ANCOVA; Difference in LS Means = -0.7, 95% CI 2-sided [-1.2 to -0.1]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.175, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-0.9 to 0.2]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.422, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-0.3 to 0.8]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.651, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.096, ANCOVA; Difference in LS Means = -0.5, 95% CI 2-sided [-1.0 to 0.1]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.860, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.511, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-0.8 to 0.4]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.286, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-0.9 to 0.3]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.004, ANCOVA; Difference in LS Means = -0.9, 95% CI 2-sided [-1.4 to -0.3]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.060, ANCOVA; Difference in LS Means = -0.5, 95% CI 2-sided [-1.1 to 0.0]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.345, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.439, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-0.7 to 0.3]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, ANCOVA; Difference in LS Means = -0.8, 95% CI 2-sided [-1.4 to 0.3]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.040, ANCOVA; Difference in LS Means = -0.6, 95% CI 2-sided [-1.1 to 0.0]

16. Secondary Outcome: Change From Baseline in UPDRS Part 2
Description: The UPDRS is a frequently used multi-item 4-part questionnaire designed to assess various aspects of Parkinson's disease severity. A total of 42 items are assessed divided across Parts 1 to 4. Part 2 assesses daily living (13 items scored from 0 [best] to 4 [worst]; total range 0-52). Assessments were obtained at baseline (predose Day 1) and 2 hours postdose at Weeks 2, 4, 6, 8, 10, and 12. For endpoint, the last postbaseline visit while on study medication was used. Change from baseline in LS means and pooled SD were obtained from an ANCOVA model with effect for treatment and baseline covariate. Negative change from baseline indicates a decrease in severity.
Time Frame: Baseline (predose Day 1) and 2 hours postdose at Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (UPDRS Part 2) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 48 | 45 | 49 | 45
Units on a Scale
  Week 2 (n=44,42,40,41,41) | 0.0 (3.13) | -1.0 (3.13) | -1.0 (3.13) | -1.2 (3.13) | 0.2 (3.13)
  Week 4 (n=40,45,41,43,43) | -0.6 (3.54) | -0.4 (3.54) | -1.8 (3.54) | -1.7 (3.54) | -0.8 (3.54)
  Week 6 (n=39,41,39,35,42) | -1.0 (3.37) | -1.3 (3.37) | -1.8 (3.37) | -0.3 (3.37) | -0.7 (3.37)
  Week 8 (n=33,42,38,37,41) | -0.2 (3.27) | -0.9 (3.27) | -2.2 (3.27) | -1.8 (3.27) | -0.9 (3.27)
  Week 10 (n=32,39,37,35,41) | -0.4 (3.63) | -0.8 (3.63) | -2.0 (3.63) | -0.8 (3.63) | -0.6 (3.63)
  Week 12 (n=31,37,36,38,37) | -0.4 (3.48) | -1.1 (3.48) | -2.7 (3.48) | -0.8 (3.48) | -0.8 (3.48)
  Endpoint (n=45,46,41,47,44) | -0.3 (3.61) | -0.9 (3.61) | -2.5 (3.61) | -0.9 (3.61) | -1.0 (3.61)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.743, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-1.1 to 1.6]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.225, ANCOVA; Difference in LS Means = -0.8, 95% CI 2-sided [-2.2 to 0.5]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.252, ANCOVA; Difference in LS Means = -0.8, 95% CI 2-sided [-2.2 to 0.6]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.173, ANCOVA; Difference in LS Means = -0.9, 95% CI 2-sided [-2.3 to 0.4]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.757, ANCOVA; Difference in LS Means = 0.2, 94% CI 2-sided [-1.3 to 1.8]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.581, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-1.1 to 1.9]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.195, ANCOVA; Difference in LS Means = -1.0, 95% CI 2-sided [-2.5 to 0.5]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.272, ANCOVA; Difference in LS Means = -0.8, 95% CI 2-sided [-2.4 to 0.7]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.758, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-1.7 to 1.2]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.416, ANCOVA; Difference in LS Means = -0.6, 95% CI 2-sided [-2.1 to 0.9]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.174, ANCOVA; Difference in LS Means = -1.0, 95% CI 2-sided [-2.5 to 0.5]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.547, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-1.1 to 2.0]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.372, ANCOVA; Difference in LS Means = 0.7, 95% CI 2-sided [-0.8 to 2.2]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.942, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-1.4 to 1.5]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.082, ANCOVA; Difference in LS Means = -1.3, 95% CI 2-sided [-2.8 to 0.2]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.267, ANCOVA; Difference in LS Means = -0.8, 95% CI 2-sided [-2.3 to 0.6]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.801, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-1.5 to 1.9]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.753, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-1.9 to 1.4]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.087, ANCOVA; Difference in LS Means = -1.4, 95% CI 2-sided [-3.1 to 0.2]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.796, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-1.9 to 1.4]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.621, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-1.3 to 2.1]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.784, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-1.8 to 1.4]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.024, ANCOVA; Difference in LS Means = -1.9, 95% CI 2-sided [-3.5 to -0.2]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.963, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-1.6 to 1.6]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.331, ANCOVA; Difference in LS Means = 0.7, 95% CI 2-sided [-0.8 to 2.3]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.898, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-1.4 to 1.6]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.058, ANCOVA; Difference in LS Means = -1.5, 95% CI 2-sided [-3.0 to 0.0]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.832, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-1.3 to 1.7]

17. Secondary Outcome: Change From Baseline in UPDRS Part 3 (1 Hour Post-dose)
Description: The UPDRS is a frequently used multi-item 4-part questionnaire designed to assess various aspects of Parkinson's disease severity. A total of 42 items are assessed divided across Parts 1 to 4. The Part 3 subscale assesses motor function across 14 categories for 27 items. Scores for each item range from 0 (best) to 4 (worst) with a total range of 0-108. Assessments were obtained at baseline (predose Day 1) and 1 hour postdose at Weeks 2, 4, 6, 8, 10, and 12. For endpoint, the last postbaseline visit while on study medication was used. Change from baseline in LS means and pooled SD were obtained from an ANCOVA model with effect for treatment and baseline covariate. Negative change from baseline indicates a decrease in severity.
Time Frame: Baseline (predose Day 1) and 1 hour postdose at Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline data (UPDRS Part 3) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 47 | 43 | 53 | 47
Units on a Scale
  Week 2 (n=42,40,37,39,43) | -1.1 (8.49) | -1.4 (8.49) | -0.9 (8.49) | -5.8 (8.49) | -2.7 (8.49)
  Week 4 (n=40,44,40,43,43) | -3.3 (8.52) | -2.4 (8.52) | -3.7 (8.52) | -5.8 (8.52) | -1.0 (8.52)
  Week 6 (n=39,41,38,33,41) | -1.2 (8.63) | -3.3 (8.63) | -3.4 (8.63) | -4.3 (8.63) | -2.4 (8.63)
  Week 8 (n=31,42,36,35,41) | -2.1 (8.82) | -2.7 (8.82) | -5.1 (8.82) | -6.8 (8.82) | -3.8 (8.82)
  Week 10 (n=31,38,36,34,41) | -2.9 (8.76) | -5.3 (8.76) | -4.1 (8.76) | -5.0 (8.76) | -1.6 (8.76)
  Week 12 (n=30,39,35,38,40) | -2.2 (9.16) | -3.3 (9.16) | -4.0 (9.16) | -5.2 (9.16) | -3.0 (9.16)
  Endpoint (n=47,47,43,53,47) | -1.9 (9.32) | -2.3 (9.32) | -3.8 (9.32) | -5.5 (9.32) | -2.2 (9.32)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.365, ANCOVA; Difference in LS Means = 1.7, 95% CI 2-sided [-2.0 to 5.3]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.476, ANCOVA; Difference in LS Means = 1.4, 95% CI 2-sided [-2.4 to 5.1]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.343, ANCOVA; Difference in LS Means = 1.8, 95% CI 2-sided [-2.0 to 5.6]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.103, ANCOVA; Difference in LS Means = -3.1, 95% CI 2-sided [-6.8 to 0.6]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.224, ANCOVA; Difference in LS Means = -2.3, 94% CI 2-sided [-6.0 to 1.4]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.448, ANCOVA; Difference in LS Means = -1.4, 95% CI 2-sided [-5.1 to 2.2]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.154, ANCOVA; Difference in LS Means = -2.7, 95% CI 2-sided [-6.4 to 1.0]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.010, ANCOVA; Difference in LS Means = -4.8, 95% CI 2-sided [-8.5 to -1.1]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.540, ANCOVA; Difference in LS Means = 1.2, 95% CI 2-sided [-2.6 to 5.0]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.646, ANCOVA; Difference in LS Means = -0.9, 95% CI 2-sided [-4.7 to 2.9]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.608, ANCOVA; Difference in LS Means = -1.0, 95% CI 2-sided [-4.9 to 2.9]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.343, ANCOVA; Difference in LS Means = -1.9, 95% CI 2-sided [-6.0 to 2.1]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.419, ANCOVA; Difference in LS Means = 1.7, 95% CI 2-sided [-2.5 to 5.9]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.562, ANCOVA; Difference in LS Means = 1.1, 95% CI 2-sided [-2.8 to 5.1]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.525, ANCOVA; Difference in LS Means = -1.3, 95% CI 2-sided [-5.3 to 2.7]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.148, ANCOVA; Difference in LS Means = -3.0, 95% CI 2-sided [-7.0 to 1.1]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.546, ANCOVA; Difference in LS Means = -1.3, 95% CI 2-sided [-5.4 to 2.9]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.068, ANCOVA; Difference in LS Means = -3.7, 95% CI 2-sided [-7.6 to 0.3]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.208, ANCOVA; Difference in LS Means = -2.5, 95% CI 2-sided [-6.5 to 1.4]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.099, ANCOVA; Difference in LS Means = -3.4, 95% CI 2-sided [-7.5 to 0.6]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.731, ANCOVA; Difference in LS Means = 0.8, 95% CI 2-sided [-3.6 to 5.1]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.861, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-4.5 to 3.8]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.621, ANCOVA; Difference in LS Means = -1.0, 95% CI 2-sided [-5.2 to 3.1]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.288, ANCOVA; Difference in LS Means = -2.2, 95% CI 2-sided [-6.4 to 1.9]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.861, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-3.5 to 4.1]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.954, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-4.0 to 3.7]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.419, ANCOVA; Difference in LS Means = -1.6, 95% CI 2-sided [-5.5 to 2.3]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.088, ANCOVA; Difference in LS Means = -3.2, 95% CI 2-sided [-6.9 to 0.5]

18. Secondary Outcome: Change From Baseline in UPDRS Part 3 (2 Hours Post-dose)
Description: The UPDRS is a frequently used multi-item 4-part questionnaire designed to assess various aspects of Parkinson's disease severity. A total of 42 items are assessed divided across Parts 1 to 4. The Part 3 subscale assesses motor function across 14 categories for 27 items. Scores for each item range from 0 (best) to 4 (worst) with a total range of 0-108. Assessments were obtained at baseline (predose Day 1) and 2 hours postdose at Weeks 2, 4, 6, 8, 10, and 12. For endpoint, the last postbaseline visit while on study medication was used. Change from baseline in LS means and pooled standard deviation were obtained from an ANCOVA model with effect for treatment and baseline covariate. Negative change from baseline indicates a decrease in severity.
Time Frame: Baseline (predose Day 1) and 2 hours postdose at Weeks 2, 4, 6, 8, 10, 12
Population: as for outcome 17
Measure: Least Squares Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 47 | 47 | 43 | 53 | 47
Units on a Scale
  Week 2 (n=44,44,41,44,44) | -2.7 (8.04) | -2.9 (8.04) | -3.5 (8.04) | -5.1 (8.04) | -2.6 (8.04)
  Week 4 (n=40,45,41,43,43) | -3.2 (8.48) | -1.5 (8.48) | -4.0 (8.48) | -6.0 (8.48) | -2.9 (8.48)
  Week 6 (n=38,41,39,34,42) | -2.5 (8.31) | -2.4 (8.31) | -4.0 (8.31) | -6.4 (8.31) | -2.5 (8.31)
  Week 8 (n=33,42,38,37,41) | -1.9 (8.85) | -1.7 (8.85) | -5.7 (8.85) | -6.9 (8.85) | -5.6 (8.85)
  Week 10 (n=32,39,37,35,41) | -3.5 (8.40) | -4.3 (8.40) | -5.2 (8.40) | -5.6 (8.40) | -3.4 (8.40)
  Week 12 (n=31,39,36,39,40) | -2.7 (8.84) | -3.1 (8.84) | -7.3 (8.84) | -6.8 (8.84) | -4.5 (8.84)
  Endpoint (n=47,47,43,53,47) | -3.0 (9.09) | -2.8 (9.09) | -5.9 (9.09) | -6.3 (9.09) | -3.1 (9.09)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.924, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-3.5 to 3.2]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.840, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-3.8 to 3.1]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.599, ANCOVA; Difference in LS Means = -0.9, 95% CI 2-sided [-4.4 to 2.5]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.134, ANCOVA; Difference in LS Means = -2.6, 95% CI 2-sided [-6.0 to 0.8]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.846, ANCOVA; Difference in LS Means = -0.4, 94% CI 2-sided [-4.1 to 3.3]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.467, ANCOVA; Difference in LS Means = 1.3, 95% CI 2-sided [-2.3 to 5.0]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.533, ANCOVA; Difference in LS Means = -1.2, 95% CI 2-sided [-4.8 to 2.5]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.094, ANCOVA; Difference in LS Means = -3.1, 95% CI 2-sided [-6.7 to 0.5]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.994, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-3.7 to 3.7]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.944, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-3.5 to 3.8]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.424, ANCOVA; Difference in LS Means = -1.5, 95% CI 2-sided [-5.1 to 2.2]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.042, ANCOVA; Difference in LS Means = -4.0, 95% CI 2-sided [-7.8 to -0.2]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.075, ANCOVA; Difference in LS Means = 3.7, 95% CI 2-sided [-0.4 to 7.8]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.052, ANCOVA; Difference in LS Means = 3.9, 95% CI 2-sided [0.0 to 7.8]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.975, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-4.0 to 3.9]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.541, ANCOVA; Difference in LS Means = -1.2, 95% CI 2-sided [-5.2 to 2.8]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.931, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-4.1 to 3.7]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.618, ANCOVA; Difference in LS Means = -1.0, 95% CI 2-sided [-4.7 to 2.8]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.341, ANCOVA; Difference in LS Means = -1.8, 95% CI 2-sided [-5.6 to 1.9]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.256, ANCOVA; Difference in LS Means = -2.2, 95% CI 2-sided [-6.0 to 1.6]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.399, ANCOVA; Difference in LS Means = 1.8, 95% CI 2-sided [-2.4 to 6.0]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.477, ANCOVA; Difference in LS Means = 1.4, 95% CI 2-sided [-2.5 to 5.4]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.172, ANCOVA; Difference in LS Means = -2.8, 95% CI 2-sided [-6.8 to 1.2]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.254, ANCOVA; Difference in LS Means = -2.3, 95% CI 2-sided [-6.2 to 1.7]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.972, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-3.6 to 3.8]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.891, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-3.5 to 4.0]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.143, ANCOVA; Difference in LS Means = -2.8, 95% CI 2-sided [-6.6 to 1.0]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.083, ANCOVA; Difference in LS Means = -3.2, 95% CI 2-sided [-6.8 to 0.4]

19. Secondary Outcome: Change From Baseline in UPDRS Part 4
Description: The UPDRS is a frequently used multi-item 4-part questionnaire designed to assess various aspects of Parkinson's disease severity. A total of 42 items are assessed divided across Parts 1 to 4. The Part 4 subscale assesses complications of therapy over the past week for a total of eleven question items. The first three questions and question 8 are rated from 0 (best) to 4 (worst), and the remaining seven questions are simple no (0) / yes (1) questions. The total subscale score ranges from 0 to 23. Assessments were obtained at baseline (predose Day 1) and 2 hours postdose at Weeks 2, 4, 6, 8, 10, and 12. For endpoint, the last postbaseline visit while on study medication was used. Change from baseline in LS means and pooled SD were obtained from an ANCOVA model with effect for treatment and baseline covariate. Negative change from baseline indicates a decrease in severity.
Time Frame: Baseline (predose Day 1) and 2 hours postdose at Weeks 2, 4, 6, 8, 10, 12
Population: The Efficacy Population consisting of all treated participants who had post-baseline date (UPDRS Part 4) for the assessment week was used for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Number analyzed (Participants) | 45 | 46 | 41 | 47 | 44
Units on a Scale
  Week 2 (n=44,42,40,41,41) | -0.3 (1.62) | -0.5 (1.62) | -0.4 (1.62) | -0.5 (1.62) | -0.8 (1.62)
  Week 4 (n=40,45,41,43,43) | -0.4 (1.71) | -0.8 (1.71) | -0.4 (1.71) | -0.5 (1.71) | -0.3 (1.71)
  Week 6 (n=39,41,39,35,42) | -0.8 (1.75) | -0.4 (1.75) | -0.3 (1.75) | -0.2 (1.75) | -0.7 (1.75)
  Week 8 (n=33,42,38,37,41) | -0.7 (2.07) | -0.8 (2.07) | -1.0 (2.07) | -0.1 (2.07) | -0.8 (2.07)
  Week 10 (n=32,39,37,35,41) | -0.8 (1.95) | -0.4 (1.95) | -0.7 (1.95) | -0.6 (1.95) | -0.3 (1.95)
  Week 12 (n=31,37,36,38,37) | -1.1 (2.05) | 0.0 (2.05) | -1.2 (2.05) | -0.7 (2.05) | -0.9 (2.05)
  Endpoint (n=45,46,41,47,44) | -0.8 (1.95) | -0.4 (1.95) | -0.8 (1.95) | -0.7 (1.95) | -0.9 (1.95)
Statistical Analysis 1: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.154, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.2 to 1.2]
Statistical Analysis 2: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.380, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.4 to 1.0]
Statistical Analysis 3: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.288, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.3 to 1.1]
Statistical Analysis 4: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.355, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.4 to 1.0]
Statistical Analysis 5: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.831, ANCOVA; Difference in LS Means = -0.1, 94% CI 2-sided [-0.8 to 0.7]
Statistical Analysis 6: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.198, ANCOVA; Difference in LS Means = -0.5, 95% CI 2-sided [-1.2 to 0.2]
Statistical Analysis 7: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.792, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-0.8 to 0.6]
Statistical Analysis 8: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.749, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-0.8 to 0.6]
Statistical Analysis 9: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.896, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-0.8 to 0.7]
Statistical Analysis 10: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.480, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.5 to 1.0]
Statistical Analysis 11: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.285, ANCOVA; Difference in LS Means = 0.4, 95% CI 2-sided [-0.4 to 1.2]
Statistical Analysis 12: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.212, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.3 to 1.3]
Statistical Analysis 13: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.883, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.9 to 1.0]
Statistical Analysis 14: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.947, ANCOVA; Difference in LS Means = 0.0, 95% CI 2-sided [-0.9 to 0.9]
Statistical Analysis 15: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.663, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-1.1 to 0.7]
Statistical Analysis 16: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.157, ANCOVA; Difference in LS Means = 0.7, 95% CI 2-sided [-0.3 to 1.6]
Statistical Analysis 17: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.283, ANCOVA; Difference in LS Means = -0.5, 95% CI 2-sided [-1.4 to 0.4]
Statistical Analysis 18: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.768, ANCOVA; Difference in LS Means = -0.1, 95% CI 2-sided [-1.0 to 0.7]
Statistical Analysis 19: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.334, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-1.3 to 0.4]
Statistical Analysis 20: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.465, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-1.2 to 0.6]
Statistical Analysis 21: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.688, ANCOVA; Difference in LS Means = -0.2, 95% CI 2-sided [-1.2 to 0.8]
Statistical Analysis 22: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.062, ANCOVA; Difference in LS Means = 0.9, 95% CI 2-sided [0.0 to 1.8]
Statistical Analysis 23: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.579, ANCOVA; Difference in LS Means = -0.3, 95% CI 2-sided [-1.2 to 0.7]
Statistical Analysis 24: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.644, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-0.7 to 1.2]
Statistical Analysis 25: Comparison: Preladenant 1 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.825, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.8 to 1.0]
Statistical Analysis 26: Comparison: Preladenant 2 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.233, ANCOVA; Difference in LS Means = 0.5, 95% CI 2-sided [-0.3 to 1.4]
Statistical Analysis 27: Comparison: Preladenant 5 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.853, ANCOVA; Difference in LS Means = 0.1, 95% CI 2-sided [-0.8 to 1.0]
Statistical Analysis 28: Comparison: Preladenant 10 mg BID vs Placebo BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.592, ANCOVA; Difference in LS Means = 0.2, 95% CI 2-sided [-0.6 to 1.1]

ADVERSE EVENTS:
Time Frame: Up to 18 weeks
Description: The Safety Population consisted of all participants who received at least one dose of study medication (either preladenant or placebo).
Arm/Group | Preladenant 1 mg BID | Preladenant 2 mg BID | Preladenant 5 mg BID | Preladenant 10 mg BID | Placebo BID
Serious Adverse Events (participants affected / at risk) | 4/49 | 2/49 | 1/47 | 3/54 | 2/47
Other Adverse Events (participants affected / at risk) | 30/49 | 29/49 | 34/47 | 37/54 | 30/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 1 mg BID (N=49) | Preladenant 2 mg BID (N=49) | Preladenant 5 mg BID (N=47) | Preladenant 10 mg BID (N=54) | Placebo BID (N=47)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SICK SINUS SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONDITION AGGRAVATED (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 1 mg BID (N=49) | Preladenant 2 mg BID (N=49) | Preladenant 5 mg BID (N=47) | Preladenant 10 mg BID (N=54) | Placebo BID (N=47)
CONSTIPATION (Gastrointestinal disorders) | 6 (7) | 1 (1) | 6 (6) | 2 (2) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 5 (7) | 4 (5) | 6 (6) | 2 (2) | 5 (5)
ASTHENIA (General disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 3 (4) | 1 (1) | 3 (3) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (2)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
FALL (Injury, poisoning and procedural complications) | 4 (4) | 4 (17) | 3 (3) | 3 (3) | 6 (11)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
C-REACTIVE PROTEIN INCREASED (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (5) | 3 (3) | 2 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 4 (4) | 3 (3) | 6 (7) | 1 (1)
DYSKINESIA (Nervous system disorders) | 4 (6) | 3 (3) | 4 (4) | 7 (8) | 6 (6)
DYSTONIA (Nervous system disorders) | 0 (0) | 1 (3) | 3 (3) | 2 (2) | 1 (2)
HEADACHE (Nervous system disorders) | 5 (10) | 2 (2) | 4 (4) | 3 (3) | 4 (4)
PARKINSON'S DISEASE (Nervous system disorders) | 5 (5) | 3 (3) | 5 (7) | 8 (9) | 3 (4)
SOMNOLENCE (Nervous system disorders) | 5 (6) | 4 (5) | 4 (4) | 7 (7) | 3 (4)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
INSOMNIA (Psychiatric disorders) | 3 (3) | 3 (4) | 4 (4) | 5 (5) | 4 (4)
HOT FLUSH (Vascular disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 2 (2) | 3 (4) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.